CLINICAL TRIAL: NCT06592703
Title: Allogenic Adipose Tissue-derived Mesenchymal Stromal Cells for the Treatment of Primary Progressive Multiple Sclerosis: an Open-label Phase I Clinical Trial.
Brief Title: Allogenic Adipose Tissue-derived Mesenchymal Stromal Cells for the Treatment of Primary Progressive Multiple Sclerosis
Acronym: MAESTRO-4MS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35RC21_9806_MAESTRO-4MS
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient (Experimental): repeated allogenic ASCs IT injections
  Interventions: Drug: Adipose tissue-derived Mesenchymal Stromal Cells

INTERVENTIONS:
Drug: Adipose tissue-derived Mesenchymal Stromal Cells — repeated allogenic ASCs IT injections

SUMMARY:
In this study, we propose, for the first time, to test the safety and the potential efficacy of repeated allogenic Adipose tissue-derived Mesenchymal Stromal Cells IT injections in Primary Progressive Multiple Sclerosis patients.

DETAILED DESCRIPTION:
In this study, the investigators propose, for the first time, to test the safety and the potential efficacy of repeated allogenic Adipose tissue-derived Mesenchymal Stromal Cells (ASCs) IT injections in Primary Progressive Multiple Sclerosis (PPMS) patients. In fact, even if autologous Bone Marrow-Mesenchymal Stromal Cells (BM-MSC) and ASCs have already been infused intrathecally in multiple sclerosis, repeated injections of allogenic ASCs have never been tested in this disease. The use of allogenic cells is driven by recent publications reporting decreased suppressive properties of autologous MSC from MS patients.

The hypothesis is that 3 repeated intrathecal (IT) injections of allogenic ASCs every 3 months will be safe and can lower disease progression in PPMS patients.

Preamble of infusing ASCs in the first patient, it's necessary to constitute and characterize the ASC bank. ASC will be obtained from Allogeneic human mesenchymal stromal cells derived from adipose tissue of a living donor.

Once the bank is available, MS patients will be screened and included in Rennes university hospital to received ASC's infusions.

MS patients will be followed for one year after inclusion

ELIGIBILITY:
Inclusion Criteria:

* Patient with Primary Progressive MS according to the criteria of Mc Donald 2017 (Thompson et al Lancet neurol, 2017)
* Age between 18 and 55 years
* EDSS score: 3 to 6 at inclusion
* Documented evidence of disability progression independent of relapse activity at any point in time over the 2 years prior to the screening visit
* Positive CSF with oligoclonal bands
* For women of childbearing potential (WOCBP), effective contraception as per the CFTG recommendations (version 1.1)
* Having signed a free, informed and written consent
* Affiliated to social security scheme

Exclusion Criteria:

* Inflammatory activity during the past year (relapses or new T2 MRI lesions)
* Disease Modifying Drugs during the past year
* Treatment with high dose corticosteroids during the 30 days preceding the inclusion
* Contra indication to lumbar puncture/intrathecal infusion: intracranial hypertension, puncture site infections, severe thrombocytopenia (<50 G/L), anticoagulant or fibrinolytic treatment
* Participation in another therapeutic trial in the last 6 months
* Adults under legal protection (safeguard of justice, curatorship, guardianship), persons deprived of their liberty, pregnant or breastfeeding women, minors, persons unable to express their consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients experiencing at least one adverse effect | 48 weeks
  Percentage of patients experiencing at least one adverse effect (AE) due to ASC infusion qualified as CTCAE V5 grade ≥ 3 or qualified as "serious" AE using the MeDRA terminology, and occurring between the first infusion and the end of the follow-up. The severity of the AE and the causality of the ASC infusion will be validated by a DSMB

SECONDARY OUTCOMES:
Description of Adverse events related to experimental product | 48 weeks
  Number and description of AE (related to the experimental product) using MedDRA terminology and CTCAE V5 at each time point during the study
Clinical disease evolution at Week24 and Week48 after treatment : Confirmed Disability Progression using Expanded Disability Status Scale score | 3 months
  Percentage of patients with 3-months Confirmed Disability Progression (CDP) between W0 and W24-W48. Disability progression will be defined as an increase of 1pt Expanded Disability Status Scale (EDSS).
  The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. It is widely used in clinical trials and in the assessment of people with MS.
  (Disability progression will be defined as an increase of 1.5 pt if baseline EDSS=0, 1pt EDSS (if baseline 1 ≤ EDSS<6), or an increase of 0.5pt if baseline EDSS is ≥ 6; confirmed at 6 months.) EDSS : Minimum Score 1, Maximum score 10, higher scores mean a worse outcome.
Clinical disease evolution at Week24 and Week48 after treatment : Expanded Disability Status Scale score | 48 weeks
  Mean change in EDSS score between W0 and W24-W48. Expanded Disability Status Scale (EDSS). The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. It is widely used in clinical trials and in the assessment of people with MS.(Disability progression will be defined as an increase of 1.5 pt if baseline EDSS=0, 1pt EDSS (if baseline 1 ≤ EDSS<6), or an increase of 0.5pt if baseline EDSS is ≥ 6; confirmed at 6 months.) EDSS : Minimum Score 1, Maximum score 10, higher scores mean a worse outcome.
Clinical disease evolution at Week24 and Week48 after treatment : Expanded Disability Status Scale score | 48 weeks
  Percentage of patients with No Evidence of Progression (NEP): Evidence of Progression is defined by (1) EDSS progression confirmed at 3 months,
  The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. It is widely used in clinical trials and in the assessment of people with MS.
  EDSS : Minimum Score 1, Maximum score 10, higher scores mean a worse outcome.
Clinical disease evolution at Week24 and Week48 after treatment : no evidence progression using 9HPT test | 48 weeks
  Percentage of patients with No Evidence of Progression (NEP): Evidence of Progression is defined by increase of at least 20% in the 9-Hole Peg Test -9HPT.
  9HPT Nine-Hole Peg Test It is a quantitative measure of hand function and is tested with the nine-hole peg test. The patient is instructed to arrange pegs into nine holes in a board by both dominant and non-dominant hands in two consecutive trials for each hand. The amount of time (in seconds) required to place and remove all nine pegs is recorded for each trial.
Clinical disease evolution at Week24 and Week48 after treatment : no evidence progression using T25-FW | 48 weeks
  Percentage of patients with No Evidence of Progression (NEP): Evidence of Progression is defined by increase of at least 20% in the Timed-25 Foot Walk -T25W
  T25W Timed 25-foot walk test (T25W) The timed 25-foot walk test (T25W) is a quantitative measure of ambulation. The T25W is a reliable test for patients with more severe gait impairment because it primarily assesses walking speed. The patient is instructed to walk a distance of 25 feet as quickly as possible. Both ends are marked with prominent signs. Note, if the patient requires his/her assistive device while walking. As the patient completes trail 1 he/she is instructed to walk back to the starting point. The time will be recorded in seconds in both trials. Time limit = 180 seconds (3 minutes). Discontinued = Patient is unable to complete a trial in 3 minutes or completes the first trial but cannot complete trial 2 after a 5-minute rest period.
Clinical disease evolution at Week24 and Week48 after treatment : MSFC mean changes | 48 weeks
  Mean change in MSFC composite score ((include -T25W, -9HPT- and PASAT-3)
  The Multiple Sclerosis Functional Composite (MSFC) was designed by "The National MS Society's Clinical Outcome Assessment Task" and is a standardized tool used to quantify the degree of disability in patients with multiple sclerosis (MS)
Quality of life disease evolution at Week24 and Week48 after treatment : Multiple Sclerosis International Quality Of Life (MusiQoL) questionnaire | 48 weeks
  Change in the MusiQOL score
  The MusiQoL is a specific questionnaire comprising 31 questions describing nine dimensions of quality of life (Appendix 1):
  activities of daily living (eight items); psychological well-being (four); relationships with friends (four); symptoms (three); relationships with family (three); relationships with the health care system (three); emotional and sexual life (two); coping (two); rejection (two).
  Each item is scored from 1 (never/not at all) to 5 (always/very much). Before calculating the score of the dimensions, the scores of negatively written items are reversed. The score of a dimension is obtained by averaging the scores of its constituent items. The dimension scores are then transformed linearly into scores ranging from 0 to 100 (100 being the maximum quality of life level). A global quality of life score is also available.
Immunophenotyping | 48 weeks
  Immunophenotyping in cerebrospinal fluid (CSF) and in blood assessing immunological and biomarkers modifications (at Week 0, Week 4, Week 12, Week 16, Week 24, Week 28, Week 48) immunophenotyping evaluation by : CSF and blood immune cells phenotyping CSF and blood cytokines and chemokines dosage MS biomarkers levels in blood and CSF (including Nfl and GFAP)
Detection of donor specific anti-HLA antibodies in the blood | 28 weeks
  Alloimmunization in blood (at Week 0, Week 4, Week 12, Week 16, Week 24, Week 28): Detection of donor specific anti-HLA antibodies in the blood
MRI parameters : gadolinium (Gd) enhancing lesions | 48 weeks
  Mean number of Gadolinium-enhancing lesions on spinal cord and cerebral MRI (Between W0 and W24-W48 and between W24- W48)
MRI parameters : new T2 lesions | 48 weeks
  Mean number of new T2 lesions on spinal cord and cerebral MRI (Between W0 and W24-W48 and between W24- W48)
MRI parameters : change in brain volume | 48 weeks
  Mean change in brain volume on cerebral MRI (Between W0 and W24-W48 and between W24- W48)
MRI parameters : change in spinal cord volume | 48 weeks
  Mean change in spinal cord volume on spinal cord MRI (Between W0 and W24-W48 and between W24- W48)

CONTACTS AND LOCATIONS:
Overall Officials: Laure MICHEL, Pr, Principal Investigator — CHU Rennes
Locations (2):
- France (2):
  - APHP Henri Mondor, Créteil
  - CHU Rennes, Rennes

IPD SHARING:
Plan to Share IPD: Undecided